CLINICAL TRIAL: NCT00942747
Title: Phase 2 Study of Temsirolimus in Refractory and Recurrent Primary CNS Lymphoma
Brief Title: Temsirolimus in Recurrent Primary Central Nervous System (CNS) Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, PD Dr. Agnieszka Korfel, PD Dr. Agnieszka Korfel, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TemPCNSL; EudraCT 2009-011277-33
Record Dates: First submitted 2009-07-20; First posted 2009-07-21 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Recurrent or Refractory Primary CNS Lymphoma
Keywords: temsirolimus, primary CNS lymphoma, PCNSL, salvage treatment
MeSH Terms: conditions — Recurrence | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temsirolimus (Experimental): Weekly IV temsirolimus
  Interventions: Drug: temsirolimus

INTERVENTIONS:
Drug: temsirolimus — Weekly infusion of 25mg Temsirolimus (first 3 patients) or 75mg Temsirolimus (all other patients) up to a maximum of 12 months in the case of continuing response to treatment
  Other Names: Torisel; CCI-770

SUMMARY:
This is an open-label trial investigating the efficacy of temsirolimus in recurrent or refractory primary CNS lymphoma (PCNSL) after initial chemotherapy with a high-dose methotrexate containing regimen. 37 patients are planned to be treated with weekly infusions of 25mg Temsirolimus (first 3 patients) or 75mg Temsirolimus (all other patients) up to a maximum of 12 months. The trial is designed in two stages, if less than one of the first 12 patients responds to treatment, the trial is stopped. In addition to efficacy, safety and penetration of temsirolimus into the cerebrospinal fluid will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Primary CNS lymphoma diagnosed histologically or by cerebrospinal fluid cytology; absence of systemic lymphoma manifestations
* Relapse or lymphoma progression after/during high-dose methotrexate containing first-line chemotherapy or alternative therapy in the case of contraindications against high-dose methotrexate
* ECOG performance score ≤ 2
* Age ≥18 years and ≤ 75 years
* Life expectancy of at least 3 months
* Absence of active infection
* Negative HIV serology
* Adequate renal function (GFR >30ml/h)
* Adequate bone marrow reserve (neutrophils > 1500/µl, platelets > 80,000/µl)
* Bilirubin <1.5x upper limit of normal (ULN), ALT and AST <3x ULN
* At least 3 weeks interval from prior cytostatic treatment
* Negative pregnancy test
* Patient accessible for treatment and follow-up
* Patient compliance
* Signed informed consent

Exclusion Criteria:

* Secondary CNS lymphoma
* Primary intraocular lymphoma
* Patient eligible for high-dose chemotherapy and autologous stem-cell transplantation
* Concurrent treatment within another clinical trial
* Concurrent other malignant disease
* Symptomatic congestive heart failure (≥NYHA II)
* Active or uncontrolled chronic infection
* Severe concomitant disease incompatible with study conduct
* History of cerebral bleeding
* Concomitant treatment with strong CYP3A4/5-inductors or -inhibitors
* Premenopausal women without highly effective contraception (defined as Pearl index <1)
* Pregnant or lactating women
* Refusal to record and pass on pseudonymized disease and treatment related data as part of the treatment protocol
* Concurrent admission to a psychiatric institution by public order

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2009-07; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Weeks 4, 12, every 12 weeks thereafter

SECONDARY OUTCOMES:
Safety | continuous
Time to progression of disease | Weeks 4, 12, every 12 weeks thereafter or upon clinical suspicion of disease progression
Penetration of temsirolimus into cerebrospinal fluid | Weeks 1, 4 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Korfel, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (6):
- Germany (6):
  - Charité Campus Benjamin Franklin, Berlin
  - Neurology, Knappschaftskrankenhaus Bochum, Bochum University, Bochum
  - Neurology, University Hospital Bonn, Bonn
  - Hematology, Klinikum Frankfurt/Oder, Frankfurt (Oder)
  - Hematology, University Hospital Heidelberg, Heidelberg
  - Klinikum Grosshadern, University Hospital Munich, Munich

REFERENCES:
- [Background] Kuhn JG, Chang SM, Wen PY, Cloughesy TF, Greenberg H, Schiff D, Conrad C, Fink KL, Robins HI, Mehta M, DeAngelis L, Raizer J, Hess K, Lamborn KR, Dancey J, Prados MD; North American Brain Tumor Consortium and the National Cancer Institute. Pharmacokinetic and tumor distribution characteristics of temsirolimus in patients with recurrent malignant glioma. Clin Cancer Res. 2007 Dec 15;13(24):7401-6. doi: 10.1158/1078-0432.CCR-07-0781. PMID 18094423
- [Background] Smith SM, Pro B, Cisneros A, Smith S, Stiff P, Lester E, Modi S, Dancey JE, Vokes EE, van Besien E. Activity of single agent temsirolimus (CCI-779) in non-mantle cell non-Hodgkin lymphoma subtypes. J Clin Oncol 2008:26 (May 20 suppl; abstr 8514).
- [Background] Hess G, Herbrecht R, Romaguera J, Verhoef G, Crump M, Gisselbrecht C, Laurell A, Offner F, Strahs A, Berkenblit A, Hanushevsky O, Clancy J, Hewes B, Moore L, Coiffier B. Phase III study to evaluate temsirolimus compared with investigator's choice therapy for the treatment of relapsed or refractory mantle cell lymphoma. J Clin Oncol. 2009 Aug 10;27(23):3822-9. doi: 10.1200/JCO.2008.20.7977. Epub 2009 Jul 6. PMID 19581539
- [Background] Ansell SM, Inwards DJ, Rowland KM Jr, Flynn PJ, Morton RF, Moore DF Jr, Kaufmann SH, Ghobrial I, Kurtin PJ, Maurer M, Allmer C, Witzig TE. Low-dose, single-agent temsirolimus for relapsed mantle cell lymphoma: a phase 2 trial in the North Central Cancer Treatment Group. Cancer. 2008 Aug 1;113(3):508-14. doi: 10.1002/cncr.23580. PMID 18543327
- [Background] Witzig TE, Geyer SM, Ghobrial I, Inwards DJ, Fonseca R, Kurtin P, Ansell SM, Luyun R, Flynn PJ, Morton RF, Dakhil SR, Gross H, Kaufmann SH. Phase II trial of single-agent temsirolimus (CCI-779) for relapsed mantle cell lymphoma. J Clin Oncol. 2005 Aug 10;23(23):5347-56. doi: 10.1200/JCO.2005.13.466. Epub 2005 Jun 27. PMID 15983389
- [Background] Costa LJ. Aspects of mTOR biology and the use of mTOR inhibitors in non-Hodgkin's lymphoma. Cancer Treat Rev. 2007 Feb;33(1):78-84. doi: 10.1016/j.ctrv.2006.10.004. Epub 2006 Dec 11. PMID 17161912
- [Derived] Korfel A, Schlegel U, Herrlinger U, Dreyling M, Schmidt C, von Baumgarten L, Pezzutto A, Grobosch T, Kebir S, Thiel E, Martus P, Kiewe P. Phase II Trial of Temsirolimus for Relapsed/Refractory Primary CNS Lymphoma. J Clin Oncol. 2016 May 20;34(15):1757-63. doi: 10.1200/JCO.2015.64.9897. Epub 2016 Mar 14. PMID 26976424